CLINICAL TRIAL: NCT02804516
Title: Recognition and Management of Early Mobilization in ICUs : Practice Patterns in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, Southeast University, China, Southeast University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 218.94.112.98/Login.aspx
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Early Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the nurse did early mobilization (Experimental): the nurses know and do what is the early mobilization in ICU
  Interventions: Behavioral: the nurse did early mobilization
- the nurse do not do early mobilization (Experimental): the nurses do not know and do what is the early mobilization in ICU
  Interventions: Behavioral: the nurse do not do early mobilization

INTERVENTIONS:
Behavioral: the nurse did early mobilization — the nurses know and do what is the early mobilization in ICU
  Arms: the nurse did early mobilization
Behavioral: the nurse do not do early mobilization — the nurses do not know and do what is the early mobilization in ICU
  Arms: the nurse do not do early mobilization

SUMMARY:
Despite evidence to support early mobilization（EM）for critically ill patients,current status in Chinese ICUs is unknown.Understanding current practice patterns and challenges is essential to inform future research and strategies.

DETAILED DESCRIPTION:
Practice guideline recommend EM in ICU,feasibility, safety and efficacy are confirmed by evidence-based data.However,the prevalence of EM in ICU patients is still low.Moreover,most of the prevalence studies come from developed countries, such as: Australia and New England the United States and Europe. Many ICUs in non-western countries are suffering from a lack of medical resources including health care personnel and medical equipment.

A retrospective observational study.To access the implementation of Chinese intensive care units and hospitals to early mobilization.Secondary objectives were to evaluate structure and process parameters of Chinese hospitals that were associated with implementation.

ELIGIBILITY:
Inclusion Criteria:Participating ICUs at least six beds ,they could be medical ,surgical or mixed

-

Exclusion Criteria:

* pediatric ICUs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
the implementation rates for early mobility | within the first 2 to 5 days of critically illness or injury
  the application of physical activity within the first 2 to 5 days of critically illness or injury

IPD SHARING:
Plan to Share IPD: Undecided